CLINICAL TRIAL: NCT01894867
Title: Magnesium Deficiency in Cirrhotic Patients
Brief Title: Magnesium in Liver Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMC13247-12CTIL
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-06

CONDITIONS: LIVER CIRRHOSIS
Keywords: LIVER CIRRHOSIS; MAGNESIUM; MINIMAL ENCEPHALOPATHY; MUSCLE WEAKNESS
MeSH Terms: conditions — Liver Cirrhosis; Muscle Weakness | interventions — Magnesium; Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- magnesium (Experimental): will get magnesium for 6 weeks
  Interventions: Dietary Supplement: magnesium
- placebo (Placebo Comparator): will get placebo for 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: magnesium — supply magnesium oxide for 6 weeks
  Other Names: magnesium oxide
  Arms: magnesium
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
Several studies have shown in patients magnesium deficiency with liver cirrhosis.

Patients with liver cirrhosis showed considerably reduced muscle strength and muscle magnesium.

We suggest addition of magnesium to patients with established cirrhosis in order to reduce the neuromuscular and neuropsychiatric manifestations of chronic liver disease.

DETAILED DESCRIPTION:
Magnesium is the fourth most abundant cation in the body and plays an important physiological role in many of its functions.

There are no readily available and easy methods to assess magnesium status but it is estimated that magnesium deficiency is a common problem.

Magnesium deficiency can cause a wide variety of features including hypocalcaemia, hypokalaemia and cardiac and neurological manifestations. Chronic low magnesium state has been associated with a number of chronic diseases including diabetes, hypertension, coronary heart disease, and osteoporosis.

There are not enough studies on magnesium status in chronic cirrhotics who may be in depletion. However , several studies have shown in patients magnesium deficiency with liver cirrhosis. Patients with liver cirrhosis showed considerably reduced muscle strength and muscle Mg . Magnesium may have a role in the neuromuscular and neuropsychiatric manifestations of chronic liver disease (hepatic encephalopathy and muscle cramps).

The use of magnesium as a therapeutic agent in asthma, myocardial infarction, and pre-eclampsia is also discussed. We suggest addition of magnesium to patients with established cirrhosis in order to reduce the neuromuscular and neuropsychiatric manifestations of chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with liver cirrhosis

Exclusion Criteria:

* pregnant women
* Patients with acute or chronic renal failure (cr>1.5)
* Congestive heart failure NYHA 3-4
* Patient with active cancer
* Patients with dementia or mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
change in minimal hepatic encephalopathy | 6 weeks

SECONDARY OUTCOMES:
change in muscle weakness | 6 weeks after intervention

OTHER OUTCOMES:
chang in other cirrhosis parameters | 6 weeks after intervention
  change in liver function test (AST ALT GPT GGT ALBUMIN INR) change in magnesium level

CONTACTS AND LOCATIONS:
Overall Officials: keren cohen, MD, Principal Investigator — Meir Medical Center
Locations (1):
- liver outpatients clinic, Meir medical center, Kfar Saba, Israel, Israel